CLINICAL TRIAL: NCT05961774
Title: The Investigation of Underlying Mechanism of Lumbar Multifidus Muscle Activation Deficits in Adults With Chronic Low Back Pain
Brief Title: The Investigation of Underlying Mechanism of Lumbar Multifidus Muscle Activation Deficits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Peemongkon Wattananon, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU-CIRB 2023/027.1503
Record Dates: First submitted 2023-07-13; First posted 2023-07-27 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Low Back Pain
Keywords: Low back pain; Transcranial magnetic stimulation; Neuromuscular electrical stimulation; Cortical excitability; Muscle activation
MeSH Terms: conditions — Low Back Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High frequency repetitive transcranial magnetic stimulation (Experimental): This group will receive high frequency repetitive transcranial magnetic stimulation.
  Interventions: Device: Transcranial magnetic stimulation
- Neuromuscular electrical stimulation (Active Comparator): This group will receive neuromuscular electrical stimulation.
  Interventions: Device: Neuromuscular electrical stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — The stimulation point is the lumbar multifidus hotspot. The parameters will be set at frequency 10 Hz, 50 number of pulses, 40 train of stimulation (5 seconds stimulation and 25 seconds inter-stimulation interval). The position of coil will be placed tangentially at 45 degrees on the LM hotspot. The stimulation will be 20 minutes.
  Arms: High frequency repetitive transcranial magnetic stimulation
Device: Neuromuscular electrical stimulation — The neuromuscular electrical stimulation will be set as interferential current 6000 Hz, amplitude 20-50 Hz with scanning mode, duration 20 minutes, intensity to elicit the LM contraction.
  Arms: Neuromuscular electrical stimulation

SUMMARY:
The goal of this clinical trial is to investigate mechanism underlying lumbar multifidus muscle (LM) activation deficits in adults with chronic low back pain (CLBP). The main questions it aim to answer is whether motor cortex or muscular level is the underlying mechanism responsible for the LM activation deficits.

Participants will:

* Undergo cortical excitability measurement using transcranial magnetic stimulation, LM activation measurement using ultrasound imaging, and force measurement using hand-held dynamometer.
* Be randomly assigned to either repetitive magnetic stimulation (rTMS) or neuromuscular electrical stimulation (NMES)
* Undergo all measurement at post-intervention Researchers will compare within and between groups to see changes in cortical excitability, LM activation, and force.

DETAILED DESCRIPTION:
Procedure The study will use a sample of convenience. The subject with CLBP will be recruited by the flyers posted at physical therapy clinic, as well as words of mouths. The participants who are interested in the study will undergo screening process for eligibility using the inclusion-exclusion criteria checklist. If the participants meet the eligibility criteria, participants will receive the brief information of the study and the consent process will be performed.

After receiving the informed consents, all participants will be requested to fill out the information sheet for demographic and clinical data. The participants will be asked to change the cloth of the top to be able to expose the lower back region. After collecting demographic and clinical data, 3-condition of LM thickness and cross-sectional area will be measured including 1) resting condition (Rest), maximum voluntary isometric contraction condition (MVIC), and maximum voluntary isometric contraction combined with neuromuscular electrical stimulation (COMB). The landmarks will be identified while the participants lay down in prone position. The landmarks include 1) lumbar spinous process of L2-L5 and 2) L4-5 facet joint (2 cm lateral to lower half of spinous process of L4). Rehabilitative ultrasound imaging (RUSI) will be used to measure LM activation and hand-held dynamometer will be used to measure force in this study across 3 conditions.

The participant will have 10 minutes rest before the transcranial magnetic stimulation (TMS). A pair of surface electrodes (Ag/AgCl, 10 mm) will be place according to SENIAM recommendation. The common ground electrode will be placed at the iliac crest. Two surface EMG electrodes will be placed relative to L4-5 along with the line joining from posterosuperior iliac spine and L1-L2 vertebral interspace (24) on the side of pain. The researcher will determine the hotspot of lumbar multifidus muscle area on the brain. The hotspot of the LM will be determined by least intensity of TMS which at least elicits 50 percent of measurable motor evoked potential (MEP) and this intensity will be the active motor threshold (AMT) of the participants. After the AMT is achieved, the 120% of AMT will be used as the intensity to induce the MEP. The MEP will be used to represent cortical excitability.

After the baseline RUSI and TMS data collection, the participants will be randomly assigned in to 2 groups include 1) NMES and high-frequency repetitive TMS (HF-rTMS) group. For HF-rTMS group, the participants will be in sitting position feet placed firmly on the floor. The stimulation point is the LM hot spot which is pre-determined by single pulse TMS as aforementioned. The HF-rTMS will be applied for participant individually. According to the theory, HF-rTMS results in facilitation of the targeted area; therefore, it will increase the excitability of the LM hot spot and potentially increase LM's neural drive and activation. The parameters will be set at frequency 10 Hz, 50 number of pulses, 40 train of stimulation (5 seconds stimulation and 25 seconds inter-stimulation interval) (34). The stimulation will approximately 20 minutes. The position of coil will be placed tangentially at 45 degrees on the LM hotspot. For the neuromuscular electrical stimulation (NMES) group, participants will be lying in prone position. The landmarks and electrodes placements are the same as mentioned in MVIC combined with NMES and LM thickness measurement. NMES parameters are interferential current 6000 Hz, amplitude 20-50 Hz with scanning mode, duration 20-minute, intensity to elicit the LM contraction (6). After the participants completed receiving the stimulation, the participant will undergo the collecting the LM thickness and force again using the same protocol.

Data will be used to 1) identify changes in cortical excitability, LM activation and force before and after stimulation at cortical level by HF-rTMS, 2) identify changes in cortical excitability, LM activation and force before and after stimulation at muscular level by NMES, and 3) compare the percent changes in cortical excitability, LM activation and force between stimulation at cortical (by HF-rTMS) and muscular (by NMES) levels.

ELIGIBILITY:
Inclusion Criteria:

* Male and female age between 18 and 40 years.
* Experience of low back pain at least 3 months, or recurrent of back pain for at least two episodes in 6 months that interferes with activities of daily living.

Exclusion Criteria:

* Spondylolysis, spondylolisthesis, spine tumor and malignancy
* Radiculopathy or myelopathy
* History of lumbar or abdominal surgery
* Pregnancy
* Neurological Disease (e.g., stroke, Parkinson, traumatic brain injury, spinal cord injury)
* Major cardiovascular diseases (e.g., heart failure, coronary artery diseases, angina pain)
* Skin lesion (e.g., skin laceration) on site of stimulation.
* Experience of lumbar motor control exercise more than or equal to 2 weeks
* Metal implantation sensitive to magnetic field, or cardiac implantations
* BMI greater or equal to 30 kg/m2
* Taking any medications that would interfere with brain stimulation (e.g., Calcium channel blockers, Na+ channel blocker, NMDA antagonist, Glutamate receptor antagonist, nicotine uptake)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Resting motor threshold | Change from baseline after 1 session
  The stimulus intensity that causes a minimum motor response in a resting muscle during single transcranial magnetic stimulation (TMS) pulses applied over the motor hotspot.
Active motor threshold | Change from baseline after 1 session
  The lowest stimulus intensity to elicit a motor evoked potential ≥ 200μV in 5 out of 10 consecutive trials during an isometric contraction of 10% maximum voluntary contraction in the target muscle.
Motor evoked potential | Change from baseline after 1 session
  The electrical signals recorded from the descending motor pathways or from muscles following stimulation of motor pathways within the brain.
Cortical silent period | Change from baseline after 1 session
  The temporary interruption of electromyographic signal from a muscle following a motor evoked potential triggered by transcranial magnetic stimulation over the primary motor cortex.
Muscle thickness | Change from baseline after 1 session
  Muscle contractility.
Muscle cross-sectional area | Change from baseline after 1 session
  Cross-sectional area can be related to joint torque production and isokinetic strength in different muscle groups.
Muscle pennation angle | Change from baseline after 1 session
  Pennation angle can represent the maximum force developed by a muscle

SECONDARY OUTCOMES:
Force generation | Change from baseline after 1 session
  Hand-held dynamometer will be used to measure muscle force.

CONTACTS AND LOCATIONS:
Overall Officials: Peemongkon Wattananon, PhD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Unidentifiable data can be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After June 2023 for 5 years.
Access Criteria: Written request will be reviewed by principal investigator.

REFERENCES:
- [Background] Songjaroen S, Sungnak P, Piriyaprasarth P, Wang HK, Laskin JJ, Wattananon P. Combined neuromuscular electrical stimulation with motor control exercise can improve lumbar multifidus activation in individuals with recurrent low back pain. Sci Rep. 2021 Jul 20;11(1):14815. doi: 10.1038/s41598-021-94402-2. PMID 34285318
- [Background] Wattananon P, Sungnak P, Songjaroen S, Kantha P, Hsu WL, Wang HK. Using neuromuscular electrical stimulation in conjunction with ultrasound imaging technique to investigate lumbar multifidus muscle activation deficit. Musculoskelet Sci Pract. 2020 Dec;50:102215. doi: 10.1016/j.msksp.2020.102215. Epub 2020 Jul 13. PMID 33220931
- [Background] Hodges PW, Danneels L. Changes in Structure and Function of the Back Muscles in Low Back Pain: Different Time Points, Observations, and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):464-476. doi: 10.2519/jospt.2019.8827. PMID 31151377
- [Background] Wallwork TL, Stanton WR, Freke M, Hides JA. The effect of chronic low back pain on size and contraction of the lumbar multifidus muscle. Man Ther. 2009 Oct;14(5):496-500. doi: 10.1016/j.math.2008.09.006. Epub 2008 Nov 21. PMID 19027343
- [Background] Tsao H, Danneels LA, Hodges PW. ISSLS prize winner: Smudging the motor brain in young adults with recurrent low back pain. Spine (Phila Pa 1976). 2011 Oct 1;36(21):1721-7. doi: 10.1097/BRS.0b013e31821c4267. PMID 21508892
- [Background] Wand BM, Parkitny L, O'Connell NE, Luomajoki H, McAuley JH, Thacker M, Moseley GL. Cortical changes in chronic low back pain: current state of the art and implications for clinical practice. Man Ther. 2011 Feb;16(1):15-20. doi: 10.1016/j.math.2010.06.008. Epub 2010 Jul 23. PMID 20655796
- [Background] Masse-Alarie H, Beaulieu LD, Preuss R, Schneider C. Corticomotor control of lumbar multifidus muscles is impaired in chronic low back pain: concurrent evidence from ultrasound imaging and double-pulse transcranial magnetic stimulation. Exp Brain Res. 2016 Apr;234(4):1033-45. doi: 10.1007/s00221-015-4528-x. Epub 2015 Dec 26. PMID 26708518
- [Background] van Dieen JH, Reeves NP, Kawchuk G, van Dillen LR, Hodges PW. Motor Control Changes in Low Back Pain: Divergence in Presentations and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):370-379. doi: 10.2519/jospt.2019.7917. Epub 2018 Jun 12. PMID 29895230
- [Background] Strutton PH, Theodorou S, Catley M, McGregor AH, Davey NJ. Corticospinal excitability in patients with chronic low back pain. J Spinal Disord Tech. 2005 Oct;18(5):420-4. doi: 10.1097/01.bsd.0000169063.84628.fe. PMID 16189454
- [Background] Masse-Alarie H, Beaulieu LD, Preuss R, Schneider C. The side of chronic low back pain matters: evidence from the primary motor cortex excitability and the postural adjustments of multifidi muscles. Exp Brain Res. 2017 Mar;235(3):647-659. doi: 10.1007/s00221-016-4834-y. Epub 2016 Nov 15. PMID 27847987
- [Background] Patricio P, Roy JS, Macedo L, Roy M, Leonard G, Hodges P, Masse-Alarie H. Repetitive transcranial magnetic stimulation alone and in combination with motor control exercise for the treatment of individuals with chronic non-specific low back pain (ExTraStim trial): study protocol for a randomised controlled trial. BMJ Open. 2021 Mar 24;11(3):e045504. doi: 10.1136/bmjopen-2020-045504. PMID 33762244
- [Background] O'Connell NE, Wand BM, Marston L, Spencer S, Desouza LH. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2014 Apr 11;(4):CD008208. doi: 10.1002/14651858.CD008208.pub3. PMID 24729198